CLINICAL TRIAL: NCT00132665
Title: Randomized Controlled Trial to Evaluate Standard Thoracic Radiotherapy With or Without Concurrent Daily Low-dose Carboplatine in Elderly Patients With Locally Advanced Non-small Cell Lung Cancer (JCOG0301, NCSLC-Elderly-CBDCA-RT Phase III)
Brief Title: Trial to Evaluate Radiotherapy With or Without CBDCA in Elderly Patients With Non-Small Cell Lung Cancer (JCOG0301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG0301; C000000059 (Registry Identifier: UMIN-CTR)
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: non-small cell lung cancer; elderly patients; carboplatin; chemoradiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Procedure/Surgery: A: Radiotherapy alone
  Interventions: Procedure: A: Radiotherapy alone
- 2 (Experimental): Drug: B: CBDCA and Radiotherapy
  Interventions: Drug: B: CBDCA and Radiotherapy

INTERVENTIONS:
Procedure: A: Radiotherapy alone — Procedure/Surgery: A: Radiotherapy alone
  Arms: 1
Drug: B: CBDCA and Radiotherapy — Drug: B: CBDCA and Radiotherapy
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate whether radiotherapy with carboplatin will result in longer survival than radiotherapy alone in elderly patients with unresectable stage III NSCLC.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether radiotherapy with carboplatin will result in longer survival than radiotherapy alone in elderly patients with unresectable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven NSCLC
* Unresectable disease
* Stage IIIA except T3N1M0 and IIIB which does not have disease extended to any contralateral hilar nodes, atelectasis of the entire lung or malignant pleural effusions
* A required radiation field of less than one half of one lung
* Measurable disease
* No previous chemotherapy or radiotherapy
* Age >= 71
* Unable to receive cisplatin-based combination chemotherapy
* ECOG performance status (PS) of 0-2
* Adequate bone marrow, lung, hepatic, and renal function
* Written informed consent

Exclusion Criteria:

* Active infection, diarrhea, ileus, uncontrolled diabetes, myocardial infarction within three months, or severe other comorbidity
* Synchronous cancer or metachronous (within 5 years) malignancy
* Interstitial pneumonia or active lung fibrosis on chest X-ray
* Severe chronic obstructive pulmonary disease, chronic bronchitis, or bronchial asthma
* Pleural or pericardial effusion
* A history of severe hypersensitivity
* Mental disorder
* Judging of inappropriate condition for this study by physician

Min Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2003-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | During the study conduct

SECONDARY OUTCOMES:
Response rate | During the study conduct
Adverse events | During the study conduct
Progression-free survival | During the study conduct
Pattern of progression/relapse | During the study conduct

CONTACTS AND LOCATIONS:
Overall Officials: Masaaki Kawahawa, MD, Study Chair — Kinki-Chuo Chest Medical Center
Locations (37):
- Japan (37):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Aichi Cancer Center,Aichi Hospital, Okazaki, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Natsuyama, Ehime
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Gifu Municipal Hospital, Gifu, Gifu
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - National Nishigunma Hospital, Shibukawa, Gunma
  - National Hospital Organization, Dohoku National Hospital, Asahikawa, Hokkaido
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Medical Center for Adults, Akashi, Hyōgo
  - Kobe City General Hospital, Kobe, Hyōgo
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Ibaraki Kenritsu Chuo Hospital & Cancer Center, Nishi-ibarakigun, Ibaraki
  - Yokohama Mucipical Citizen's Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kumamoto Regional Medical Center Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Okayama, Okayama-ken
  - Osaka Prefectural Medical Center for Respiratory and Allergic Disease, Habikino, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka, Osaka
  - Graduate School of Medicine, Osaka City University, Osaka, Osaka
  - Osaka General Medical Center, Osaka, Osaka
  - Kinki University School of Medicine, Ōsaka-sayama, Osaka
  - Kinki-Chuo Chest Medical Center, Sakai, Osaka
  - National Hospital Organization Toneyama National Hospital, Toyonaka, Osaka
  - Saitama Cancer Center, Kita-adachi, Saitama
  - Sizuoka Cancer Center, Sunto-gun, Shizuoka
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital, Koto-ku, Tokyo
  - Toranomon Hospital, Minato-ku, Tokyo
  - International Medical Center of Japan, Shinjuku-ku, Tokyo
  - Yamagata Prefectural Central Hospital, Yamagata, Yamagata

REFERENCES:
- [Derived] Atagi S, Mizusawa J, Ishikura S, Takahashi T, Okamoto H, Tanaka H, Goto K, Nakagawa K, Harada M, Takeda Y, Nogami N, Fujita Y, Kasai T, Kishi K, Sawa T, Takeda K, Tomii K, Satouchi M, Seto T, Ohe Y. Chemoradiotherapy in Elderly Patients With Non-Small-Cell Lung Cancer: Long-Term Follow-Up of a Randomized Trial (JCOG0301). Clin Lung Cancer. 2018 Sep;19(5):e619-e627. doi: 10.1016/j.cllc.2018.04.018. Epub 2018 May 5. PMID 29887243
- [Derived] Atagi S, Kawahara M, Yokoyama A, Okamoto H, Yamamoto N, Ohe Y, Sawa T, Ishikura S, Shibata T, Fukuda H, Saijo N, Tamura T; Japan Clinical Oncology Group Lung Cancer Study Group. Thoracic radiotherapy with or without daily low-dose carboplatin in elderly patients with non-small-cell lung cancer: a randomised, controlled, phase 3 trial by the Japan Clinical Oncology Group (JCOG0301). Lancet Oncol. 2012 Jul;13(7):671-8. doi: 10.1016/S1470-2045(12)70139-0. Epub 2012 May 22. PMID 22622008
- See also: Related Info — http://www.jcog.jp/